CLINICAL TRIAL: NCT04296097
Title: Evaluation of Deep Brain Stimulation (DBS) of the Right Operculum 3 (OP3) in Permanent Non-pulsatile Disabling Tinnitus (TINNOP3-DBS)
Acronym: TINNOP3-DBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government); Équipe 5 Neuroimagerie et perfusion cérébrale, Grenoble Institut des Neurosciences (GIN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 38RC18.208; 2019-A01562-55 (Other: ANSM ID RCB)
Record Dates: First submitted 2020-02-24; First posted 2020-03-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Severe Permanent Uni or Bilateral Non-pulsatile Tinnitus; Without Associated Vestibular Pathology; Resistant to Therapeutic Failure; With or Without Hearing Loss
Keywords: Tinnitus; Deep Brain Stimulation (DBS); Right operculum 3 (OP3); Functional Magnetic Resonance Imaging (fMRI); Magnetoencephalography (MEG); Local Field Potential (LFP); Visual Analog Scale (VAS); Tinnitus Handicap Inventory (THI) questionnaire; Hospital Anxiety and Depression Scale (HAD); Cross-over study; Double blind design
MeSH Terms: conditions — Tinnitus; Depression

STUDY DESIGN:
Intervention Model Description: Deep Brain Stimulation (DBS) of the parieto-insular region at the level of the right operculum 3 (OP3)
Who Masked: Participant, Investigator
Masking Description: Crossover study conducted in double blind design :
  * one month Deep Brain Stimulation (DBS) ON, 15 days wash out stimulation OFF, and one month Deep Brain Stimulation (DBS) OFF or
  * one month Deep Brain Stimulation (DBS) OFF, 15 days wash out stimulation OFF, and one month Deep Brain Stimulation (DBS) ON
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep Brain Stimulation (DBS) activated (Experimental): Patients with severe permanent non-pulsatile tinnitus treated by Deep Brain Stimulation (DBS) in position ON
  Interventions: Device: DBS
- Deep Brain Stimulation (DBS) non-activated (Other): Patients with severe permanent non-pulsatile tinnitus treated by Deep Brain Stimulation (DBS) in position OFF
  Interventions: Device: DBS

INTERVENTIONS:
Device: DBS — Deep Brain Stimulation (DBS) of the parieto-insular region at the level of the right operculum 3 (OP3)

SUMMARY:
This pilot study aims at evaluating the effectiveness of the treatment of unilateral or bilateral, non-pulsatile, disabling, tinnitus, without vestibular dysfunction, using Deep Brain Stimulation (DBS) of the parieto-insular right operculum 3 (OP3) in a cross-over, double study design.

DETAILED DESCRIPTION:
Subjective, non-pulsatile, permanent, severe, tinnitus, refractory to all treatment are very disabling. They can lead to serious depression and suicidal behavior, which justifies the development of innovative therapeutic options. Current management is essentially based on psychological therapy and / or prosthetic, to improve for hearing loss that can be frequently associated. In fact, the main objective is habituation for these patients, but when the tinnitus is too intense, it is impossible. Three recent publications in functional magnetic resonance imaging (fMRI) have reported a novel physiopathological hypothesis to explain the appearance of subjective tinnitus. They highlight the prominent role of the right operculum 3 (OP3), a deep opercular region (parieto-insular junction) in the emergence of this symptom. The investigators hypothesize that inhibition of this region using high frequency stimulation could, significantly improve the intensity of the symptom and consequently their quality of life in this selected population.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years old,
2. Uni or bilateral permanent non-pulsatile tinnitus, without associated vestibular pathology, with or without hearing loss,
3. Severe tinnitus resistant to treatment failure,
4. Tinnitus intensity on the Visual Analog Scale (VAS) ≥ 7,
5. Presenting a quality of life score on the Tinnitus Handicap Inventory (THI) questionnaire> 76 (= grade 5),
6. Social security affiliates or beneficiaries of such a scheme
7. Informed and written consent signed by the patient.

Exclusion Criteria:

1. Vestibular dysfunction (balance disorder),
2. Epilepsy,
3. Intercurrent serious pathology,
4. Brain tumor,
5. Contraindication to surgery or anesthesia,
6. History of cerebral infection with herpesvirus,
7. With a contraindication to the practice of MRI, MEG, Computerized Tomography (CT) scan,
8. Under anticoagulants and antiaggregants (Anti vitamin K, low molecular weight heparin, aspirin and derivatives, clopidogrel antiplatelet agents and assimilated, new oral anticoagulants (NACO)) for which a therapeutic window can not be opened within 3 months before and after the surgery,
9. Included in another therapeutic protocol,
10. Progressive dementia or psychiatric illness,
11. Presenting a suicidal risk deemed important for less than 3 months (Montgomery and Asberg depression scale (MADRS): suicidality item (item 10) score> 2),
12. Enforced hospitalisation,
13. Pregnant, parturient or breastfeeding, lack of contraception in patients with the capacity to procreate,
14. Subject to a legal protection measure,
15. Deprived of liberty by judicial or administrative decision,
16. Isolated patient without any contact in case of emergency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the treatment using Deep Brain Stimulation (DBS) of the right operculum 3 (OP3). | 2.5 months
  Difference in intensity of tinnitus Visual Analog Scale (VAS) [0/10 : higher scores mean better outcome] between the end and the beginning of each of the two periods of the crossover.

SECONDARY OUTCOMES:
Incidence of DBS Treatment on Emergent Adverse Events (Tolerance) after surgical intervention and stimulation following the implantation of the DBS medical device. | 15 months
  Emergent Adverse events (partial or general epileptic seizures, worsening of tinnitus, surgical complications, ...): 1) post-operative computed tomography (CT); 2) Clinical evaluation.
Evaluation of the subjective effect of stimulation on quality of life. | 15 months
  Scores on the Tinnitus Handicap Inventory (THI) questionnaire [0/100 : higher scores mean worse outcome] at 6 months (early phase) and at 15 months compared to the preoperative THI of the same patient.
Evaluation of the subjective effect of stimulation on anxiety / depression. | 15 months
  Scores on the Hospital Anxiety and Depression Scale (HAD) [0/21 : higher scores mean worse outcome] at 6 months (early phase) and at 15 months compared to preoperative HAD of the same patient.
Changes comparison of the connectivity of OP3 explored by functional Magnetic Resonance Imaging (fMRI) at 1.5 T. | 15 months
  Functional Magnetic Resonance Imaging records (fMRI 1.5 T) performed preoperatively and at 15 months postoperatively.
Connectivities changes of the right OP3 measured by magnetoencephalography (MEG) at baseline 'preoperatively) and the post op (within 1 week) and at long term follow up (15 months) with active stimulation (ON) and inactive (OFF) during MEG recording. | 15 months
  Magnetoencephalography (MEG) records at baseline (preoperatively) and the post op (within 1 week) and at long term follow up (15 months) with active stimulation (ON) and inactive (OFF) during MEG recording.
Characterization of the Local Field Potential (LFP) recorded and correlations with tinnitus features perceived by the patient, based on their intensity and characteristic. | One week
  Local Field Potential (LFP) records on the electrode when the patient perceives tinnitus features 1) intraoperatively 2) before the implantation of the stimulator.

CONTACTS AND LOCATIONS:
Locations (1):
- CLINATEC, Grenoble, France

REFERENCES:
- [Background] Job A, Paucod JC, O'Beirne GA, Delon-Martin C. Cortical representation of tympanic membrane movements due to pressure variation: an fMRI study. Hum Brain Mapp. 2011 May;32(5):744-9. doi: 10.1002/hbm.21063. PMID 21484948
- [Background] Job A, Pons Y, Lamalle L, Jaillard A, Buck K, Segebarth C, Delon-Martin C. Abnormal cortical sensorimotor activity during "Target" sound detection in subjects with acute acoustic trauma sequelae: an fMRI study. Brain Behav. 2012 Mar;2(2):187-99. doi: 10.1002/brb3.21. PMID 22574285
- [Background] Job A, Jacob R, Pons Y, Raynal M, Kossowski M, Gauthier J, Lombard B, Delon-Martin C. Specific activation of operculum 3 (OP3) brain region during provoked tinnitus-related phantom auditory perceptions in humans. Brain Struct Funct. 2016 Mar;221(2):913-22. doi: 10.1007/s00429-014-0944-0. Epub 2014 Dec 12. PMID 25503643
- [Background] Eickhoff SB, Grefkes C, Zilles K, Fink GR. The somatotopic organization of cytoarchitectonic areas on the human parietal operculum. Cereb Cortex. 2007 Aug;17(8):1800-11. doi: 10.1093/cercor/bhl090. Epub 2006 Oct 10. PMID 17032710
- [Background] Maliia MD, Donos C, Barborica A, Popa I, Ciurea J, Cinatti S, Mindruta I. Functional mapping and effective connectivity of the human operculum. Cortex. 2018 Dec;109:303-321. doi: 10.1016/j.cortex.2018.08.024. Epub 2018 Sep 10. PMID 30414541